CLINICAL TRIAL: NCT06939920
Title: NIV With Airway Washout for Dual Limb Ventilation: Improvement in Minute Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Fisher and Paykel Healthcare
Record Dates: First submitted 2025-03-31; First posted 2025-04-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Failure Requiring Non Invasive Ventilation
Keywords: Non-invasive ventilation; OptiNIV; Airway washout
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized, non-blinded, crossover pilot investigation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visairo (Active Comparator): Visairo is a commercially available sub nasal oronasal mask that has a similar design as the interventional OptiNIV Dual Mask
  Interventions: Other: non-invasive ventilation
- OptiNIV Dual (Experimental): Like the commercially available OptiNIV mask, this mask provides NIV with airway washout but now for dual limb ventilators.
  Interventions: Other: Non-invasive ventilation mask with airway washout

INTERVENTIONS:
Other: Non-invasive ventilation mask with airway washout — Non-invasive ventilation mask with airway washout for dual limb ventilators
  Arms: OptiNIV Dual
Other: non-invasive ventilation — standard state of the art non-invasive ventilation
  Arms: Visairo

SUMMARY:
This is a prospective, non-randomized, non-blinded, crossover feasibility investigation to assess the safety, usability, and efficacy of the investigational mask in the hospital environment. Eligible patients that are stable in NIV and able to give informed consent will be approached and if they consent the patient will be included in the study. If potential participants decline, normal hospital care will be continued. The enrolled participant will receive NIV on the commercially available Visairo mask for one hour during which their ventilatory parameters will be logged. Then the participant will be switched to the investigational mask for another hour. The ventilator data will be collected for these two hours. At the end of the intervention the participant will be reverted to their original mask. The medical staff will be asked to fill out the case report form pertaining to the function and usability of the investigational mask compared to the conventional mask.

DETAILED DESCRIPTION:
In an acute setting, Non-invasive ventilation (NIV) is a method of delivering respiratory support without using an endotracheal tube. It's a first-line treatment for specific conditions like COPD exacerbations and acute cardiogenic pulmonary edema. NIV aims to improve gas exchange, reduce work of breathing, avoid intubation, and reduce complications.

For patients with COPD exacerbations and acute cardiogenic pulmonary edema NIV is a first line therapy. NIV is also considered for other conditions like acute respiratory failure due to asthma exacerbation and in immunocompromised individuals with acute respiratory insufficiency. Additionally, it can be used in post-operative respiratory failure, for difficult weaning, and to prevent post-extubation failure.

NIV has been shown to result in overall better outcomes than mechanical ventilation with reduced mortality and morbidity, fewer ICU acquired infections improved lung function and shorter ICU stays. The severity of the respiratory insufficiency influences the likelihood of successful NIV. One factor associated with respiratory sufficiency is respiratory dead space. This is the volume in the respiratory apparatus that does not partake in gas exchange and in the ventilated patient includes the volume in the equipment, the conductive airways and pathological respiratory tissue. A high dead-space fraction early in the course of the illness is association with increased risk of death.9 Particularly in patients that have a small tidal volume and high respiratory rate, or patients with an increased physiological dead space due to lung disease, a change in instrumental dead space can have a large impact on alveolar minute ventilation. Improved alveolar ventilation can improve CO2 elimination and help to reduce respiratory acidosis as well as improve oxygen delivery.10, 11 This can consequently reduce the respiratory effort required by the patient. 12 If the physician instead chooses to keep arterial CO2 concentration (PaCO2) constant, a reduction of instrumental dead space will allow a reduction of tidal volume, plateau pressure, driving pressure, or a reduction of the respiratory rate and thus a reduction in work of breathing.

NIV with washout improves ventilation compared to conventional NIV by reducing expired air in each breath. This may result in faster normalization of ventilatory gasses and a reduced work of breathing, the patient may improve more rapidly as alveolar ventilation is improved. Or, allow for a reduction in pressure for similar ventilatory benefits, potentially improving NIV tolerance and therapy adherence. In stable COPD patients, NIV with Airway Washout resulted in a significant reduction in minute ventilation compared to conventional NIV. This was approximately 19% lower with OptiNIV compared to conventional NIV.15 In this study minute ventilation will be calculated from the RR and Vt retrieved from the ventilator to asses improvement in ventilation over the study period, this feasibility pilot aims to establish efficacy of airway washout and whether the increased leak required for dead space flushing does not impact safety, usability and performance. When airway washout for dual limb ventilators becomes widely available it may improve NIV therapy efficacy by improving ventilation or reducing the pressure needed for a similar level of ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to the ICU prescribed NIV and stable
* Able to receive therapy on a sub-nasal (under-the-nose) mask
* Are 18 years old or older

Exclusion Criteria:

* Contraindicated for NIV
* NIV is likely to fail and/or intubation be required, at the medical staff's discretion
* Bilevel pressure of ≥ 30 cmH2O required
* Do not fit the investigational mask or the standard mask
* Pregnancy (tested under standard care)
* Unable to tolerate NIV for the duration of the investigation
* Agitated
* Unable to understand the consent process

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
minute ventilation | The first 5 minutes on each mask will be compared to the last 5 minutes on the same mask and the differences compared by paired T-test.
  To establish that the performance of the investigational mask is on par or better than a conventional NIV. Comparing the Visairo and the investigational masks for a reduction in minute ventilation over the 1 hour study period. We anticipate a reduction in minute ventilation that is 2L/min less than in the comparator mask. This will be established with a paired T test over the first 5 and last 5 min of data extracted from the ventilator.

SECONDARY OUTCOMES:
Ventilator data (pressure) | Ventilator data can be logged in 5 min intervals the study data ie 1h on visairo and 1h on optiniv dual will be exported to USB after the participant has concluded both arms.
  Data will be downloaded from the ventilator after the trial is concluded. This will include pressure flow and leak data as well as alarms and settings. This data will be compared between arms to see if the ventilators behave statistically different between arms and if so on what parameters. Pressure data will be compared via paired T-test between arms.
Ventilator data (flow) | Ventilator data can be logged in 5 min intervals the study data ie 1h on visairo and 1h on optiniv dual will be exported to USB after the participant has concluded both arms.
  Data will be downloaded from the ventilator after the trial is concluded. This will include pressure flow and leak data as well as alarms and settings. This data will be compared between arms to see if the ventilators behave statistically different between arms and if so on what parameters. Flow data will be compared via paired T-test between arms.
user feedback | once both arms are completed, right after the 2 hours on NIV
  To establish that the safety, usability and performance of the investigational mask is on par with a conventional NIV, according to the attending nurse/healthcare provider. The attending nurse/healthcare provider will complete a questionnaire, comparing the Visairo and the OptiNIV dual masks. Whether the masks performed similarly, ease of therapy establishment, if any asynchrony was noticed, if in their opinion the participants were equally comfortable in both masks. This is qualitative data, each of the 5 questions will be given a score from 1-5 for a maximum of 25. a Score of 8-17 being neutral below will favor the conventional mask above will favor the investigational mask.
Ventilator data (leak) | Ventilator data can be logged in 5 min intervals the study data ie 1h on visairo and 1h on optiniv dual will be exported to USB after the participant has concluded both arms.
  Data will be downloaded from the ventilator after the trial is concluded. This will include pressure flow and leak data as well as alarms and settings. This data will be compared between arms to see if the ventilators behave statistically different between arms and if so on what parameters. Leak data will be compared via paired T-test between arms.
Ventilator data (alarms) | Ventilator data can be logged in 5 min intervals the study data ie 1h on visairo and 1h on optiniv dual will be exported to USB after the participant has concluded both arms.
  Data will be downloaded from the ventilator after the trial is concluded. This will include pressure flow and leak data as well as alarms and settings. This data will be compared between arms to see if the ventilators behave statistically different between arms and if so on what parameters. Alarm data will be compared via paired T-test between arms.